CLINICAL TRIAL: NCT06148792
Title: A Revised Tafenoquine Dose to Improve Radical Cure for Vivax Malaria - TAfenoquine DOsing REvised
Brief Title: A Revised Tafenoquine Dose to Improve Radical Cure for Vivax Malaria
Acronym: TADORE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Menzies School of Health Research (Other)
Collaborators: University of Melbourne (Other); Fundação de Medicina Tropical Dr. Heitor Vieira Dourado (Other); Arba Minch University (Other); Addis Ababa University (Other); Eijkman Research Center for Molecular Biology, National Research and Innovation Agency, Indonesia (Unknown); Curtin University (Other); Papua New Guinea Institute of Medical Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TADORE
Record Dates: First submitted 2023-11-19; First posted 2023-11-28 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-04

CONDITIONS: Vivax Malaria
MeSH Terms: conditions — Malaria, Vivax | interventions — tafenoquine; Primaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- TQRevised (Experimental): Patients are treated with schizontocidal treatment plus a single weight-based oral dose of TQ (target dose 7.5mg/kg)
  Interventions: Drug: Tafenoquine
- TQStandard (Active Comparator): Patients are treated with schizontocidal treatment plus single fixed oral dose of 300mg TQ (TQStandard)
  Interventions: Drug: Tafenoquine
- PQ7 (Experimental): Patients are treated with schizontocidal treatment plus oral high dose PQ (total dose 7 mg/kg) over 7 days (PQ7)
  Interventions: Drug: Primaquine

INTERVENTIONS:
Drug: Tafenoquine — oral treatment
  Arms: TQRevised; TQStandard
Drug: Primaquine — oral treatment
  Arms: PQ7

SUMMARY:
The goal of this clinical trial is to assess the efficacy and safety or a revised weight band tafenoquine dose in vivax malaria patients. The main question[s] it aims to answer are:

* is a revised weight-based TQ regimen (TQRevised: target dose 7.5mg/kg) non-inferior to high dose primaquine (7mg/kg over 7 days)
* is a revised weight-based TQ regimen (TQRevised: target dose 7.5mg/kg) superior to fixed dose tafenoquine (300mg)
* is the tolerability and safety of TQRevised acceptable
* is TQRevised acceptable and feasible Participants will receive a tafenoquine target dose 7.5mg/kg in weight bands. Researchers will compare this to patients receiving a fixed dose tafenoquine and high dose primaquine to see if safe and effective.

ELIGIBILITY:
Inclusion Criteria:

* P. vivax peripheral parasitaemia (mono-infection)
* G6PD normal status (G6PD activity ≥70% of the adjusted male median as determined by the Standard G6PD (SDBioline, ROK))
* Fever (temperature ≥37.5⁰C) or history of fever in the preceding 48 hours
* Written informed consent
* Living in the study area and willing to be followed for six months

Exclusion Criteria:

* Danger signs or symptoms of severe malaria
* Anaemia (defined as Hb <8g/dl)
* Pregnant or lactating females
* Regular use of drugs with haemolytic potential
* Known hypersensitivity to any of the study drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1090 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
The incidence risk of vivax parasitaemia | 4 months
  The incidence risk (time to first event) of any P. vivax parasitaemia during the 4-month follow up period as determined by microscopy.
  * compared between TQRevised and the PQ7 (non-inferiority)
  * compared between TQRevised and TQStandard (superiority)

SECONDARY OUTCOMES:
The incidence risk of vivax parasitaemia | 4 months
  The incidence risk (time to first event) of any P. vivax parasitaemia during the 4-month follow up period as determined by microscopy compared between TQStandard and PQ7
The incidence risk of symptomatic vivax parasitaemia | 4 months
  The incidence risk (time to first event) of symptomatic P. vivax parasitaemia during the 4 months follow up period as determined by microscopy
The incidence risk of vivax parasitaemia | 6 months
  The incidence risk (time to first event) of any P. vivax parasitaemia at 6-month follow up as determined by microscopy
The incidence risk of symptomatic vivax parasitaemia | 6 months
  The incidence risk (time to first event) of symptomatic P. vivax parasitaemia at 6-month follow up as determined by microscopy
The incidence rate of vivax parasitaemia | 6 months
  The incidence rate (events per person-time) of any P. vivax parasitaemia during the 6 months follow up period as determined by microscopy
The incidence rate of symptomatic vivax parasitaemia | 6 months
  The incidence rate (events per person-time) of symptomatic P. vivax parasitaemia during the 6 months follow up period as determined by microscopy
The incidence risk of anaemia | 7 and 14 days, 6 months
  The incidence risk of developing severe anaemia (Hb < 5g/dl) or moderate (5g/dl and <7g/dl) anaemia within 7 and 14 days of starting treatment and/or requiring blood transfusion within the 6 months follow up period
The incidence risk of an acute drop in Hb | 7 and 14 days
  The incidence risk of an acute drop in Hb of >25% to <7g/dl within 7 and 14 days of starting treatment
Adverse events | 42 days
  The number and proportion of adverse and serious adverse events in each arm within 42 days after start of treatment
Meth Hb concentration | day 7
  day 7 methaemoglobin concentration

CONTACTS AND LOCATIONS:
Overall Officials: Kamala N Thriemer, PhD, Principal Investigator — Menzies School of Health Research
Locations (4):
- Dr Marcus Lacerda, Manaus, Brazil
- Arba Minch General Hospital, Arba Minch, Ethiopia
- Puskesmas Hanura, Hanura, Indonesia
- Dr Moses Laman and Dr Brioni Moore, Alexishafen, Papua New Guinea

IPD SHARING:
Plan to Share IPD: Yes